CLINICAL TRIAL: NCT06953973
Title: Investigation of the Effectiveness of Tecar Therapy in Patients With Chronic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Muhammed İhsan KODAK, Dr, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/369
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tecar Therapy + Standard Physiotherapy Program (Experimental)
  Interventions: Other: Tecar Therapy; Other: Standard Physiotherapy Program
- Sham Tecar Therapy + Standard Physiotherapy Program (Sham Comparator)
  Interventions: Other: Sham Tecar Therapy; Other: Standard Physiotherapy Program
- Standard Physiotherapy Program (Active Comparator)
  Interventions: Other: Standard Physiotherapy Program

INTERVENTIONS:
Other: Tecar Therapy — Tecar Therapy will be applied by a specialist physiotherapist with WINTECARE T-PLUS-Switzerland. Participants in the experimental group included in the Tecar therapy application will be applied to the muscle groups in the neck region at a fixed frequency of 0.448 Mhz for 10 minutes.
  Arms: Tecar Therapy + Standard Physiotherapy Program
Other: Sham Tecar Therapy — Tecar Therapy will be applied by a specialist physiotherapist with WINTECARE T-PLUS-Switzerland. The patient will be positioned as in the Tecar group, but the heating feature of the device will not be activated.
  Arms: Sham Tecar Therapy + Standard Physiotherapy Program
Other: Standard Physiotherapy Program — This study will include routinely applied conventional physiotherapy, heat modalities, electrotherapy (transcutaneous electrical nerve stimulation (TENS) and ultrasound therapy), and exercises. In this study, hot pack will be used to induce vasodilation and reduce muscle spasm. Hot pack will be used for 15 minutes to relax muscle spasms and increase soft tissue flexibility. TENS is a simple noninvasive modality and is widely used in both acute and chronic neck pain. In our study, 50 Hz conventional TENS with a pulse duration of <150 microseconds will be used. TENS will be applied to the painful area of the neck for 20 minutes. Ultrasound therapy used to warm deep tissues is one of the most frequently used physical therapy methods. An ultrasound device (Chattanooga, USA) will be used in the study. Ultrasound gel will be applied circularly with a thickness of 2-3 mm. Ultrasound will be applied with a 4 cm2 probe for 5 minutes with a frequency of 1 MHz and 1.5 Wt/cm2. Within the scope o

SUMMARY:
Study Design This study was planned as a randomized controlled, double-blind study. Chronic neck pain diagnosed by a specialist physician will be divided into 3 groups with a randomization model. Interested individuals will be included in the study if they meet the inclusion criteria and sign the 'Informed Voluntary Consent Form' after the study is explained.

Patients will be divided into 3 groups with a randomization (secretary not in the study) model.

Patients who choose 1 will be applied Tecar Therapy + Standard Physiotherapy Program (SFP), those who choose 2 will be applied Sham Tecar Therapy +SFP and those who choose 3 will be applied SFP. The first and last evaluations of all 3 groups will be made by the same blind evaluator.

Randomization After the study is explained to the patients with chronic neck pain who meet the inclusion and exclusion criteria, those who volunteer will be asked to sign the "Informed Voluntary Consent Form". Those who volunteer to participate in the study will be randomly assigned to Group 1, Group 2 or 3. Participants will be randomly assigned to a card. Those who draw number 1 will be assigned to the SFP+Tecar Therapy group, those who draw number 2 will be assigned to the Sham Tecar Therapy + SFP group, and those who draw number 3 will be assigned to the SFP only group.

Visual Analog Scale (VAS) The pain intensity felt by the participants in the knee joint during rest and activity will be evaluated with VAS. VAS is an easy-to-use scale as it does not have any language and is frequently applied in clinics. Individuals will be asked to describe the pain they feel during the test on a 10 cm scale as "0" (no pain) and "10" (unbearable pain). A 34% decrease in VAS after TKA is considered clinically significant.

Neck Disability Index Neck Disability Index (NDI) was developed by Vernon et al. The Turkish version study was conducted by Aslan et al. The NDI includes a total of 10 questions such as pain, personal care, concentration, work, driving, and sleeping. Each question is scored between 0 and 5 points. A score of 0 means no restriction, and a score of 50 means full restriction. A score between 0-4 indicates no restriction, a score between 5-14 indicates mild restriction, a score between 14-24 indicates moderate restriction, a score between 25-34 indicates severe restriction, and a score above 35 indicates restriction.

Tampa Kinesiophobia Scale TKÖ is a 17-question checklist and is used in acute and chronic low back pain, fibromyalgia, musculoskeletal injuries, and whiplash-related diseases. The scale uses a 4-point Likert scale (1= I strongly disagree, 4= I strongly agree). A total score is calculated after reversing items 4, 8, 12, and 16. The person receives a total score between 17-68. A high score on the scale indicates that the person has high kinesiophobia. The validity and reliability of the questionnaire in Turkish was conducted by Tunca Yılmaz et al.

Quality of Life (SF-12) SF-12 consists of 8 sub-dimensions and 12 items, including physical functioning (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functioning (1 item), emotional role (2 items) and mental health (2 items). While the items related to physical and emotional role are answered dichotomously (yes or no), other items have Likert-type options ranging from 3 to 6. The total score of the survey varies between 0-100, with higher scores representing better health. The validity and reliability of the survey in Turkish was performed by Soylu et al.

Hospital Anxiety Depression Scale The scale is used to determine the risk of anxiety and depression in patients, and to measure their levels and changes in severity. The scale consists of a total of 14 questions. Seven of these (odd numbers) measure anxiety, while the other seven (even numbers) measure depression. The scale provides a four-point Likert-type measurement. Each item is scored differently. Items 1, 3, 5, 6, 8, 10, 11 and 13 show decreasing severity and are scored in the form of 3, 2, 1, 0. On the other hand, items 2, 4, 7, 9, 12 and 14 are scored in the form of 0, 1, 2, 3. The total scores of the subscales are obtained by adding these item scores. While items 1, 3, 5, 7, 9, 11 and 13 are added for the anxiety subscale, the scores of items 2, 4, 6, 8, 10, 12 and 14 are added for the depression subscale. Each heading is scored between 0-21. High scores indicate high anxiety and depression. The Hospital Anxiety and Depression Scale was developed by Zigmond and Snaith in 1983. In our country, the validity and reliability study was conducted by Aydemir in 1997.

Global Rating Of Change Scale This scale is frequently used to evaluate patient satisfaction in orthopedic clinical studies. It is designed to determine the amount of improvement or deterioration of the patient over time. In GRC, which is a Likert-type scale, the options in the plus and minus value ranges and the labels assigned to these degrees

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-55,
* Having neck pain for 3 months or longer,
* Being able to come to the hospital for a standart physiotherapy program

Exclusion Criteria:

* Patients who have had a cervical spine injury or surgery
* Patients with neck pain secondary to a neurological or vascular disorder or neoplasia
* Patients with radiculopathy and neurological deficits
* Patients with a history of inflammatory or infective arthritis in the cervical spine
* Patients who have received a physical therapy program in the last 6 months
* Patients with open wounds or risk of infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 0-4 weeks
Neck Disability İndex | 0-4 weeks

SECONDARY OUTCOMES:
Tampa Kinesiophobia Scale | 0-4 weeks
Short Form-12 (SF-12) | 0-4 weeks
Hospital Anxiety Depression Scale | 0-4 weeks
Global Rating Of Change Scale-GRC | 0-4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No